CLINICAL TRIAL: NCT06975956
Title: Evaluation of Sexual Function and Quality of Life Tests in Patients Who Underwent Manchester Operation for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cemile ilhan, Principal investigator, Specialist Physician in Obstetrics and Gynecology, Bagcilar Training and Research Hospital
Other Study IDs: 2023/23
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: Pelvic organ prolapse; Manchester operation
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female patients who underwent Manchester operation for pelvic organ prolapse.: Complaints, demographic characteristics and gynecologic examinations of the patients who underwent Manchester operation will be performed. Preoperative and postoperative 6th month pelvic examination will include POP Q scoring, Female Sexual Function Index (FSFI) questionnaire consisting of 19 questions to evaluate sexual life, Prolapse Quality of Questionnaire (PQOL) consisting of 20 questions to evaluate quality of life.

SUMMARY:
Pelvic organ prolapse is a condition that affects sexual health and quality of life at all ages. The efficacy of the Manchester operation planned in appropriate patients and its effects on the sexual function and quality of life of the patient were investigated and it was thought that uterine preservation should be offered as a treatment option in the young age group of patients who want uterine preservation and in cases with comorbidity and short operation time required.

DETAILED DESCRIPTION:
Patients with ≥2 pelvic organ prolapse according to POP Q staging system who are examined in the urogynecology outpatient clinic with the complaint of prolapse will be presented to the gynecology council. As a result of P0P Q scoring, patients with cervical elongation findings with C point ≥0, D point ≤-4 and estimated cervical length ≥5 cm, age, fertility, patient's desire to preserve the uterus, comorbid diseases will be evaluated and patients who are planned for Manchester operation in the council decision will be included in the study. All patients will have undergone ultrasonography and cervical smear screening. Cervical, uterine and ovarian malignant pathologies will be excluded. Anamnesis information and test results of these patients who require operation will be obtained from the electronic information system of our hospital and the files of the patients. In the case report form, the patient's age, obstetric anamnesis, BMI (body mass index), POP Q scoring in preoperative and postoperative 6th month pelvic examination, Female Sexual Function Index (FSFI) questionnaire consisting of 19 questions to evaluate sexual life, Prolapse Quality of Questionnaire (P QOL) questionnaire consisting of 20 questions to evaluate quality of life will be performed. Duration of operation, estimated blood loss, postoperative hemogram change will be obtained from the operation records. Preoperative and postoperative 6th month POP Q scoring, sexual function and quality of life tests were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Manchester operation for pelvic organ prolapse

Exclusion Criteria:

* Patients who refused to participate in the study. Patients undergoing hysterectomy for pelvic organ prolapse, cancer patients, patients with uterine, cervical and ovarian malignancy.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing Manchester operation for pelvic organ prolapse
Study Population: Patients undergoing Manchester operation for pelvic organ prolapse
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Function as will be measured by the Female Sexual Function Index (FSFI) in patients undergoing Manchester operation for pelvic organ prolapse. | Preoperative and 6 months postoperative
  The FSFI is a 19-item questionnaire evaluating six domains(desire, arousal, lubrication, orgasm, sexual satisfaction and pain) of female sexual function. Total scores range from 2 to 36; higher scores reflect better sexual function
Change in Quality of Life as will be measured by Prolapse quality of life tests (PQOL) in patients undergoing Manchester operation for pelvic organ prolapse | Preoperative and 6 months postoperative
  PQOL questionnaire consists of 20 questions about general health perceptions, prolapse impact, role imitation, physical limitations, social limitation, personal relationships, emotions, sleep/energy, severity measures. Each section is scored with a minimum score of 0 and a maximum score of 100. A high total score indicates a greater impairment of quality of life.
Change in Pelvic Organ Support as will be measured by the Pelvic Organ | Preoperative and 6 months postoperative
  The POP-Q system measures vaginal point locations relative to the hymen in centimeters (e.g., Aa, Ba, C, D points). Improvement is reflected by a reduction in positive or elevated values.

CONTACTS AND LOCATIONS:
Locations (1):
- Bağcılar Training and Reserach Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Park YJ, Kong MK, Lee J, Kim EH, Bai SW. Manchester Operation: An Effective Treatment for Uterine Prolapse Caused by True Cervical Elongation. Yonsei Med J. 2019 Nov;60(11):1074-1080. doi: 10.3349/ymj.2019.60.11.1074. PMID 31637890